CLINICAL TRIAL: NCT05477134
Title: Arginine Metabolism in Pediatric Type 2 Diabetes
Brief Title: Arginine Metabolism in Youth With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mustafa Tosur, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-51936
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Children; Pediatric type 2 diabetes; Pediatric diabetes; Arginine; Youth
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study cohort consisting of youth with type 2 diabetes and healthy controls (Experimental): In Study Day 1, participants will be given a primed dose of stable isotopes followed by continuous intravenous infusions for 5 hours. The investigators will use the following isotopes: U-13C6-Arg, 5,5-2H2-Cit, 15N2-Orn, 2H5-Phe, and Na13CO3.
  On Study Day 2, participants will drink a 75-gram glucose solution prior to an oral glucose tolerance test.
  On Study Day 3, participants will drink a 75-gram glucose solution and will be injected 5-gram arginine into their veins.
  Interventions: Other: Stable isotope infusion, oral glucose ingestion, intravenous arginine bolus

INTERVENTIONS:
Other: Stable isotope infusion, oral glucose ingestion, intravenous arginine bolus — On separate study days, each participant will have a stable isotope infusion, ingest oral glucose, and be given an intravenous arginine bolus.

SUMMARY:
Type 2 diabetes (T2D), once considered only "a disease of older ages," is now a significant public health concern in youth. Although it is characterized by insulin resistance and impaired insulin secretion, its precise etiology and pathogenesis are not yet fully understood. This study aims to (1) explore arginine metabolism in youth with T2D via safe, minimally invasive kinetic experiments using stable isotope tracers and targeted metabolomics, and (2) determine the effect of exogenous arginine administration on β-cell function in youth with T2D, potentially supporting the use of this safe, low-cost, and readily available nutrient to improve pediatric diabetes outcomes.

DETAILED DESCRIPTION:
In parallel with the youth obesity epidemic, type 2 diabetes (T2D) in youth is becoming a significant public health concern. The incidence of pediatric T2D increased by 50% during the past decade, and recent data show that T2D accounts for one in four newly-diagnosed diabetes cases in children. Youth with T2D have an aggressive disease course and a rapid decline in β-cell function, and many also have multiple cardiovascular disease risk factors at an early age. The disease is characterized by insulin resistance and impaired insulin secretion, but the molecular underpinnings of T2D are not yet fully elucidated. This study aims to uncover the role of arginine metabolism in the pathogenesis of youth with T2D and the effect of exogenous arginine administration on β-cell function in them.

Arginine is a known stimulant of insulin secretion in pancreatic β-cells. Nitric oxide (NO) is synthesized from arginine by NO synthase, and arginine stimulates insulin secretion in both NO-mediated and NO-independent mechanisms by stimulating guanylate cyclase, membrane depolarization, and metabolic by-products. The effects of arginine in pancreatic β-cells are dependent on the cells' available arginine concentration. Kinetic techniques using isotope tracer infusions and targeted metabolomics provide a unique opportunity to determine "intracellular" arginine availability and its relative contribution of various pathways to this pool. Such studies in adults with T2D have shown that arginine and NO play roles in the pathogenesis of T2D by affecting insulin secretion and insulin sensitivity. In the preliminary data on children with T2D, the investigators found that children with T2D had lower fasting arginine, citrulline (arginine precursor), and glutamine (citrulline precursor) levels. In this proposal, the investigators will seek kinetic validation of these hypothesis-generating observations to investigate the role of arginine metabolism in youth with T2D. Our central hypothesis is that youth with T2D have inadequate arginine availability (Aim 1), leading to suboptimal β-cell function, which can be restored by exogenous arginine administration (Aim 2). If our hypotheses are proven, arginine supplementation will play a clinically vital role in improving diabetes outcomes in this population as a safe, low-cost, and readily available nutrient.

ELIGIBILITY:
Inclusion Criteria:

1. Youth with type 2 diabetes and healthy controls who meet other inclusion criteria outlined below.
2. Age and pubertal stage criteria (12- to 20-year-old girls who are postmenarchal, and 14- to 20-year-old boys who are at Tanner stage 5 genitalia),
3. Additional criteria for youth with diabetes: i. diagnosis of T2D, and ii. diabetes duration between 3 months and 10 years.

Exclusion Criteria:

1. Previous history of diabetic ketoacidosis (DKA)
2. Poorly controlled diabetes defined as HbA1c >7.5%,
3. Abnormal liver, thyroid, gonadal or adrenal functions,
4. Renal insufficiency defined by eGFR (estimated glomerular filtration rate) <90 mL/min/1.73 m2,
5. Any glucose lowering medications except metformin, insulin and liraglutide

(7) Any medication use that will likely to interfere amino acid metabolism, (8) Any hormonal replacement therapy, and (9) Pregnancy.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The difference in arginine availability | 1 day
  Arginine availability will be assessed and compared between youth with type 2 diabetes and healthy controls.

SECONDARY OUTCOMES:
The difference in insulin secretion and the effect of intravenous arginine bolus on insulin secretion | 1 day
  Insulin secretion will be assessed and compared between youth with type 2 diabetes and healthy controls using oral glucose tolerance tests and modified oral glucose tolerance tests including intravenous arginine administration. The effect of arginine bolus on insulin secretion will be compared between the groups.
The difference in insulin sensitivity and the effect of intravenous arginine bolus on insulin sensitivity | 1 day
  Insulin sensitivity will be assessed and compared between youth with type 2 diabetes and healthy controls using oral glucose tolerance tests and modified oral glucose tolerance tests including intravenous arginine administration. The effect of arginine bolus on insulin sensitivity will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Tosur, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital / Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No